CLINICAL TRIAL: NCT02659657
Title: Prophylaxis Roles of Low Dose of IL-2 Treatment on GVHD After Haploidentical Transplantation
Brief Title: Prophylaxis Roles of IL-2 Treatment on GVHD After Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Chief of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016PHB006-01
Record Dates: First submitted 2016-01-08; First posted 2016-01-20 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute Graft-versus-host Disease
MeSH Terms: interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin-2 interventions (Experimental): Patients with standard risk hematologic malignancies undergoing an unmodified haploidentical HCT will be eligible. Once patients achieved neutrophil engraftment will be given IL-2, 0.4×10E+6/M2/d, 3 times a week (separated by at least 1 day between injections) until day +90 (+/- 7 days).
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Interleukin-2 (IL-2), 0.4×10E+6/M2/d, 3 times a week (separated by at least 1 day between injections) until day +90 (+/- 7 days)
  Other Names: IL-2

SUMMARY:
The effects of haploidentical rhG-CSF-mobilized unmanipulated blood and marrow transplantation (HBMT) on hematological malignancies are well established.The aim of this prospective cohort trial is to determine if acute graft-versus-host disease (aGVHD) could be decreased with IL2 therapy post HBMT.

DETAILED DESCRIPTION:
The effects of haploidentical rhG-CSF-mobilized unmanipulated blood and marrow transplantation (HBMT) on hematological malignancies are well established.The aim of this prospective cohort trial is to determine if acute graft-versus-host disease (aGVHD) could be decreased with IL2 therapy post HBMT.low dose of IL-2 (40 million U/m2) will be administered from WBC engraftment to day 90 post haploidentical transplantation. IL-2 will be administered three times a week.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 15-65 years old
2. Acute leukemia in complete remission (CR1/CR2) who received myeloablative haploidentical allo-HSCT
3. WBC engraftment (ANC>500/ul for continuous 3 days)
4. At least +7d
5. Less than or equal to +15d
6. non T-ALL
7. no active II-IV aGVHD
8. no severe infections
9. Karnofsky score greater than or equal to 90%
10. Haploidentical donor from sibling, children or father
11. Ensure that informed consent signed and faxed to Research Coordinator

Exclusion Criteria:

1. Exposure to any other clinical trials prior to enrollment
2. Active malignant disease relapses or MRD positive
3. Active, uncontrolled infection
4. Inability to comply with IL-2 treatment regimen
5. Active, uncontrolled II-IV aGVHD
6. Haploidentical donor from mother or collateral donors
7. Clinical Signs of severe pulmonary dysfunction
8. Clinical Signs of sever cardiac dysfunction
9. Receiving corticosteroids as GVHD treatment

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
II-IV acute graft-versus-host disease (aGVHD) post transplantation | Day 100 post transplantation
  cumultive incidence of II-IV acute graft-versus-host disease (aGVHD) post transplantation

SECONDARY OUTCOMES:
Severe chronic GVHD post transplantation | 1 year post transplantation
  cumulative incidence of severe chronic GVHD post transplantation
CMV infection post transplantation | Day 100 post transplantation
  cumulative incidence of CMV infection post transplantation
Measureable residual disease (MRD)-positive test post transplantation | 1 year
  cumulative incidence of MRD+ post transplantation
Hematological relapse post transplantation | 1 year
  Cumulative incidence of hematological relapse post transplantation
Disease-free free survival post transplantation | 1 year
  Cumulative incidence of DFS post transplantation
Overall survival post transplantation | 1 year
  Cumulative incidence of OS post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Principal Investigator — Peking University Intitute of Hematology
Locations (1):
- Peking University Institute of Hematology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No